CLINICAL TRIAL: NCT01209494
Title: The EU TrigTreat Clinical Study: An Advanced Diagnostics and Observational Trial for Arrhythmia Risk Stratification and Correlation With Genotype
Brief Title: An Arrhythmia Risk Stratification and Genetic Trial
Acronym: EUTrigTreat
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Collaborators: UMC Utrecht (Other); KU Leuven (Other); University of Athens (Other)
Responsible Party: Principal Investigator, Markus Zabel, Associate Professor, Head of Clinical Electrophysiology, University Medical Center Goettingen
Other Study IDs: HEALTH-F2-2009-241526
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Cardiomyopathies, Primary; Arrhythmia; Sudden Cardiac Death; Calcium Metabolism Disorders
Keywords: sudden cardiac death; implantable cardioverter defibrillator; ventricular arrhythmias; genetic syndromes; calcium metabolism; ventricular repolarization; ECG; T wave; programmed electrical stimulation; alternans; late potentials; risk stratification
MeSH Terms: conditions — Cardiomyopathies; Arrhythmias, Cardiac; Death, Sudden, Cardiac; Calcium Metabolism Disorders; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood specimens for genetic analyses
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Invasive EP Study Group: 200 patients are studied before clinically indicated (according to AHA/ACC/ESC guidelines) first ICD implantation or ICD exchange. Invasive EP study is performed to test inducibility of malignant arrhythmia. In addition MAP recordings are performed for measurements of restitution properties. Pacing is done for 12-lead ECG and MAP recordings for analysis of BVR and TWA, if applicable.
- Noninvasive EP Study Group: The assignment of patients to the invasive and noninvasive EP groups does not occur by randomization or for intervention.
  In the noninvasive EP study group, 500 patients with chronically implanted ICD (>3 month after implantation) are investigated using non-invasive EP study via ICD programmer. Programmed electrical stimulation is performed to test for inducibility of malignant arrhythmia. In addition pacing is done for measurements of BVR from the 12-lead ECG.

SUMMARY:
The prospective EUTrigTreat multi-center study is an observational, advanced diagnostics and genetic risk stratification trial in patients with standard indications for ICD treatment, with and without myocardial infarction in their history.

Its aims are fourfold: 1) To accurately risk stratify a large cohort of implantable cardioverter-defibrillator (ICD) patients for ICD shock risk and mortality using traditional risk markers as well as genetic markers 2) To find a link between repolarization biomarkers and genetic markers of calcium metabolism. 3) To compare invasive and noninvasive electrophysiologic (EP) testing systematically 4) To assess temporal changes of typical noninvasive risk stratifiers and their prognostic implication.

In five European academic clinical centers, 700 ICD patients are prospectively enrolled (optionally the number of enrolled patients may be expanded to 1000 patients). Comprehensive non-invasive risk stratifying ECG diagnostics including beat-to-beat variability of repolarization (BVR) are applied, and candidate genes associated with malignant arrhythmias are analyzed. Programmed electrical stimulation is performed to test for inducibility of malignant ventricular arrhythmias and BVR. In a subset of patients, electrophysiologic studies include recording of monophasic action potentials (MAP) from the right ventricle for assessment of restitution properties. Non-invasive risk stratifying ECG methods are repeated annually. Outcome (mortality, ICD shocks) will be assessed until September 2014.

DETAILED DESCRIPTION:
An increasing number of patients receive implantable cardioverter-defibrillators for primary and secondary prevention of sudden cardiac death. Within this group, it is difficult to differentiate between patients at high risk with need for additional treatment and, on the other hand, patients at low risk without benefit from implantable cardioverter-defibrillator therapy. Risk stratification techniques have been studied extensively over the last decades, but no conclusive recommendations can be found in the current guidelines for prevention of SCD. Furthermore, new genetic markers associated with sudden cardiac death were discovered recently, however, have not been implemented in concurrent risk analysis. Last, time dependent changes of risk stratification assessment are unknown.

The prospective EUTrigTreat multi-center study is an observational, advanced diagnostics and genetic risk stratification trial in patients with standard indications for ICD treatment and without myocardial infarction in their history.

Its aims are fourfold: 1) To accurately risk stratify a large cohort of implantable cardioverter-defibrillator (ICD) patients for ICD shock risk and mortality using traditional risk markers as well as genetic markers 2) To find a link between repolarization biomarkers and genetic markers of calcium metabolism. 3) To compare invasive and noninvasive electrophysiologic (EP) testing systematically 4) To assess temporal changes of typical noninvasive risk stratifiers and their prognostic implication.

In four European academic clinical centers, 700 ICD patients are prospectively enrolled. Optionally, the number of patients may be expanded to 1000. Comprehensive non-invasive risk stratifying ECG diagnostics including beat-to-beat variability of repolarization (BVR) are applied, and candidate genes associated with malignant arrhythmias are analyzed. Programmed electrical stimulation is performed to test for inducibility of malignant ventricular arrhythmias and BVR. In a subset of patients, electrophysiologic studies include recording of monophasic action potentials (MAP) from the right ventricle for assessment of restitution properties. Non-invasive risk stratifying ECG methods are repeated annually. Outcome (mortality, ICD shocks) will be assessed until September 2014.

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for ICD treatment according to ACC/AHA/ESC guidelines for primary or secondary prevention of SCD
* Age ≥ 18 years
* Nonischemic cardiomyopathies: DCM, HCM/HOCM, ARVC or
* Channelopathies: Brugada, LQT, CPVT or
* Idiopathic VT/VF or
* Diffuse coronary artery disease, without transmural myocardial infarction in history (ACS and NSTEMI with CK maximum of 400 U/l allowed)

Exclusion Criteria:

* Unstable cardiac disease
* PCI or CABG < 3 months ago
* Implantation of a CRT device < 6 months ago
* ICD unable to deliver programmed ventricular stimulation via programmer (only in the noninvasive EP study group)
* Women of childbearing potential in case of positive pregnancy test at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard indications for ICD treatment according to ACC/AHA/ESC guidelines with and without myocardial infarction in their history are eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 672 (Actual)
Dates: Start 2010-01; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Total Mortality | 2010-2014

SECONDARY OUTCOMES:
Sudden Cardiac, Cardiac and Non-Cardiac Mortality | 2010-2014
  The standard definition of SCD applied. A cardiac death is defined as any death presumed to have occurred from a cardiac cause other than SCD. Non-cardiac deaths are all other deaths.
Appropriate and Inappropriate Shocks | 2010-2014
  Appropriate shock is a secondary endpoint. ICD shock is classified as appropriate if delivered for a true ventricular tachyarrhythmia in the VT or VF zone. Appropriate ICD shock is classified as 1 primarily delivered in the VF zone, 2 secondarily delivered as a backup to failed ATP in the VT zone or 3 secondarily delivered after acceleration of failed ATP to VF zone.
  Inappropriate shock is a secondary endpoint. Inappropriate shock is an ICD shock caused by oversensing of cardiac or non-cardiac electrical signals as VT or VF, or by inappropriate interpretation of SVT as VT/VF by the device.
Secondary Composite Endpoints | 2010-2014
  A secondary composite endpoint of total mortality and appropriate ICD shocks is defined. Another secondary composite endpoint is defined as the sum of appropriate and inappropriate ICD shocks, i.e. all ICD shocks.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zabel, M.D., Study Director — University Medical Center Goettingen; Marc A. Vos, Ph.D., Principal Investigator — UMC Utrecht; Panagotia Flevari, M.D., Principal Investigator — University of Athens; Rik Willems, M.D., Principal Investigator — KU Leuven
Locations (4):
- Katholieke Universiteit Leuven, Dept. of Cardiology, Leuven, Belgium
- University Medical Center Goettingen, Dept. of Cardiology and Pneumology, Göttingen, Germany
- Attikon Hospital University of Athens, BRFAA, Dept. of Cardiology, Athens, Greece
- Universitair Medisch Centrum Utrecht, Depts. of Cardiology and Physiology, Utrecht, Netherlands

REFERENCES:
- [Background] Koller MT, Schaer B, Wolbers M, Sticherling C, Bucher HC, Osswald S. Death without prior appropriate implantable cardioverter-defibrillator therapy: a competing risk study. Circulation. 2008 Apr 15;117(15):1918-26. doi: 10.1161/CIRCULATIONAHA.107.742155. Epub 2008 Apr 7. PMID 18391108
- [Background] Poole JE, Johnson GW, Hellkamp AS, Anderson J, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Fishbein DP, Packer DL, Mark DB, Lee KL, Bardy GH. Prognostic importance of defibrillator shocks in patients with heart failure. N Engl J Med. 2008 Sep 4;359(10):1009-17. doi: 10.1056/NEJMoa071098. PMID 18768944
- [Background] Vollmann D, Luthje L, Vonhof S, Unterberg C. Inappropriate therapy and fatal proarrhythmia by an implantable cardioverter-defibrillator. Heart Rhythm. 2005 Mar;2(3):307-9. doi: 10.1016/j.hrthm.2004.11.019. No abstract available. PMID 15851324
- [Background] Zabel M, Malik M, Hnatkova K, Papademetriou V, Pittaras A, Fletcher RD, Franz MR. Analysis of T-wave morphology from the 12-lead electrocardiogram for prediction of long-term prognosis in male US veterans. Circulation. 2002 Mar 5;105(9):1066-70. doi: 10.1161/hc0902.104598. PMID 11877356
- [Background] Zabel M, Acar B, Klingenheben T, Franz MR, Hohnloser SH, Malik M. Analysis of 12-lead T-wave morphology for risk stratification after myocardial infarction. Circulation. 2000 Sep 12;102(11):1252-7. doi: 10.1161/01.cir.102.11.1252. PMID 10982539
- [Background] Bloomfield DM, Hohnloser SH, Cohen RJ. Interpretation and classification of microvolt T wave alternans tests. J Cardiovasc Electrophysiol. 2002 May;13(5):502-12. doi: 10.1046/j.1540-8167.2002.00502.x. PMID 12030535
- [Background] Schmidt G, Malik M, Barthel P, Schneider R, Ulm K, Rolnitzky L, Camm AJ, Bigger JT Jr, Schomig A. Heart-rate turbulence after ventricular premature beats as a predictor of mortality after acute myocardial infarction. Lancet. 1999 Apr 24;353(9162):1390-6. doi: 10.1016/S0140-6736(98)08428-1. PMID 10227219
- [Background] Franz MR, Chin MC, Sharkey HR, Griffin JC, Scheinman MM. A new single catheter technique for simultaneous measurement of action potential duration and refractory period in vivo. J Am Coll Cardiol. 1990 Oct;16(4):878-86. doi: 10.1016/s0735-1097(10)80336-5. PMID 2212368
- [Background] Hummel JD, Strickberger SA, Daoud E, Niebauer M, Bakr O, Man KC, Williamson BD, Morady F. Results and efficiency of programmed ventricular stimulation with four extrastimuli compared with one, two, and three extrastimuli. Circulation. 1994 Dec;90(6):2827-32. doi: 10.1161/01.cir.90.6.2827. PMID 7994827
- [Background] Thomsen MB, Volders PG, Beekman JD, Matz J, Vos MA. Beat-to-Beat variability of repolarization determines proarrhythmic outcome in dogs susceptible to drug-induced torsades de pointes. J Am Coll Cardiol. 2006 Sep 19;48(6):1268-76. doi: 10.1016/j.jacc.2006.05.048. Epub 2006 Aug 28. PMID 16979017
- [Background] Narayan SM, Franz MR, Lalani G, Kim J, Sastry A. T-wave alternans, restitution of human action potential duration, and outcome. J Am Coll Cardiol. 2007 Dec 18;50(25):2385-92. doi: 10.1016/j.jacc.2007.10.011. PMID 18154963
- [Background] Arvanitis DA, Sanoudou D, Kolokathis F, Vafiadaki E, Papalouka V, Kontrogianni-Konstantopoulos A, Theodorakis GN, Paraskevaidis IA, Adamopoulos S, Dorn GW 2nd, Kremastinos DT, Kranias EG. The Ser96Ala variant in histidine-rich calcium-binding protein is associated with life-threatening ventricular arrhythmias in idiopathic dilated cardiomyopathy. Eur Heart J. 2008 Oct;29(20):2514-25. doi: 10.1093/eurheartj/ehn328. Epub 2008 Jul 9. PMID 18617481
- [Background] Lehnart SE, Lederer WJ. An antidote for calcium leak: targeting molecular arrhythmia mechanisms. J Mol Cell Cardiol. 2010 Feb;48(2):279-82. doi: 10.1016/j.yjmcc.2009.11.005. Epub 2009 Nov 26. No abstract available. PMID 19931542
- [Derived] Seegers J, Vos MA, Flevari P, Willems R, Sohns C, Vollmann D, Luthje L, Kremastinos DT, Flore V, Meine M, Tuinenburg A, Myles RC, Simon D, Brockmoller J, Friede T, Hasenfuss G, Lehnart SE, Zabel M; EUTrigTreat Clinical Study Investigators. Rationale, objectives, and design of the EUTrigTreat clinical study: a prospective observational study for arrhythmia risk stratification and assessment of interrelationships among repolarization markers and genotype. Europace. 2012 Mar;14(3):416-22. doi: 10.1093/europace/eur352. Epub 2011 Nov 23. PMID 22117037